CLINICAL TRIAL: NCT06094660
Title: Patients With Knee Pain Caused by Osteoarthritis: Comparison of Conservative Medical Management With RadioFrequency Ablation or Chemical Neurolysis of the Genicular Nerves With Phenol
Brief Title: RFA or Chemical Neurolysis of the Genicular Nerves Compared to Conservative Treatment for Knee Pain Caused by OA
Acronym: RADIOPHENOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dijklander Ziekenhuis (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Bravis Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOC 045
Record Dates: First submitted 2023-09-12; First posted 2023-10-23 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Osteo Arthritis Knee; Knee Pain Chronic
Keywords: Pain; Thermal ablation; Phenol neurolysis; Genicular nerve
MeSH Terms: conditions — Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chemical ablation of the genicular nerves with Phenol 6% (Active Comparator): Chemical ablation with phenol is done by injection of 1,5ml of phenol 6 % at the superomedial, the superolateral and the inferomedial genicular nerve.
  Interventions: Procedure: Diagnostic genicular nerve block; Procedure: Genicular nerve block with Phenol 6%
- Radiofrequency ablation (RFA) of the genicular nerves (Active Comparator): In our study we will make two RFA lesions at every target with 80°C for 90 seconds with a 5mm active tip. So we will make 6 lesions in total. The targets are the superomedial, the superolateral and the inferomedial genicular nerve.
  Interventions: Procedure: Diagnostic genicular nerve block; Procedure: Genicular nerve block with Radiofrequency Ablation (RFA)
- Conservative treatment (No Intervention): Examples of allowed conservative treatments during the study are patient education, physical therapy, weight loss and different pharmacological treatments.

INTERVENTIONS:
Procedure: Diagnostic genicular nerve block — Diagnostic block will be done with 1,5ml of Lidocaine 2% at the 3 target sites: the superomedial, the superolateral and the inferomedial genicular nerve.
  Arms: Chemical ablation of the genicular nerves with Phenol 6%; Radiofrequency ablation (RFA) of the genicular nerves
Procedure: Genicular nerve block with Radiofrequency Ablation (RFA) — Genicular nerve block with RFA will be performed at 3 target sites: the superomedial, the superolateral and the inferomedial genicular nerve.
  Radiofrequency ablation (RFA) is performed by creating two RFA lesions at the 3 treatment sites (6 lesions in total) after local anesthesia with 1,5ml lidocaine 2%. The lesions are made by heating the 5mm active tip of the needle to 80°C for 90 seconds.
  Arms: Radiofrequency ablation (RFA) of the genicular nerves
Procedure: Genicular nerve block with Phenol 6% — Genicular nerve block with Phenol 6% will be performed at 3 target sites: the superomedial, the superolateral and the inferomedial genicular nerve.
  Chemical ablation with phenol is done by injection of 1 ,5ml of phenol 6 % at the 3 target sites after infiltration with contrast dye to rule out intravascular injection. Because infiltration with phenol is painless, prior infiltration of the target site with al local anaesthetic is not necessary.
  Arms: Chemical ablation of the genicular nerves with Phenol 6%

SUMMARY:
A randomised controlled triall (RCT) with three parallel arms comparing the functional outcome of chemical ablation with phenol and radiofrequency ablation (RFA) of the genicular nerves with conservative treatment in patients with chronic knee pain caused by osteoarthritis (OA).

DETAILED DESCRIPTION:
In guidelines for knee osteoarthritis (OA), conservative treatments are physical therapy, analgesics and intra-articular injections with corticosteroids. In severe OA and persisting symptomatic cases the golden standard is joint replacing surgery. A less invasive technique is ablation of the sensory (genicular) nerves of the knee. This technique is beneficial for younger patients as a bridge to surgery or patients that cannot undergo total knee arthroplasty (TKA) due to comorbid health conditions. Nerve ablation can either be done with chemical agents or thermal energy.

Although there are numerous studies on genicular nerve block for chronic knee pain caused by OA, there are just a few small studies that compare genicular nerve block with conservative treatment.To be able to determine if genicular nerve ablation is efficacious to serve the gap between conservative treatment and TKA, this randomised controlled trial (RCT) compares two forms of genicular nerve ablation (radiofrequency and phenolisation; intervention) with conservative treatment (control) up to 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of both sexes, >35 years who are not a candidate for TKA due to young age, old age, comorbidity or technical reasons.
2. OKS < 30 on a scale from 0 (severe function) to 48 points (satisfactory function).
3. Continued pain in the target knee that is moderate to severe (defined as NRS ≥ 6 on an 11-point NRS scale) either constantly or with motion despite at least 3 months of conservative treatments. Conservative treatment can include: active physiotherapy, pharmacological treatment of pain (acetaminophen or NSAIDs) and intra-articular corticosteroid infiltration.
4. Radiologic confirmation of arthritis for the target knee. Defined as the Kellgren Lawrence (KL) score of 2 or more on X-ray or MRI.

Exclusion Criteria:

1. Patient with prior ablation of the genicular nerves, prior partial, resurfacing, or TKA of the target knee (residual hardware).
2. Patient with a history of neurovascular injury or recent trauma of the lower extremities.
3. Patient with chronic widespread pain.
4. Polyneuropathy and/or radicular pain in the lower extremities.
5. Patient is currently implanted with a neurostimulator.
6. Local or systemic infection (bacteraemia).
7. Uncontrolled immune suppression.
8. Intra-articular injections (steroids, hyaluronic acid, platelet enriched plasma, stem cell, …) in the target knee within 90 days from randomisation.
9. Arthroscopic debridement/lavage into the target knee within 180 days from randomisation.
10. BMI<18,5 kg/m2 and patients with minimal subcutaneous tissue thickness that would not accommodate ablation with phenol or radio frequency (risk of skin burns).
11. Allergies to products used during the procedure (lidocaine, phenol, contrast dye).
12. Patients who have a planned TKA in the near future, defined as patients who already have agreed on a date for the TKA procedure.
13. Patients with psychosocial problems as determined by the investigator.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Knee function measured with the Oxford Knee score (OKS) | During intake, before the intervention or study start in conservative group (T=0) and during the follow up visits (T=1 at 6weeks, T=2 at 3 months, T=3 at 6 months and T=4 at 12 months after the intervention or study start).
  Questionnaire with 12 items. Scores can range from 0 to 48, with 48 being the best outcome and a lower score indicates more functional limitations and pain.

SECONDARY OUTCOMES:
Osteoartritis (OA) measured by the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Before the intervention or study start in conservative group (T=0) and during the follow up visits (T=1 at 6weeks, T=2 at 3 months, T=3 at 6 months and T=4 at 12 months after the intervention or study start).
  We will use the WOMAC in the Likert version where question are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. So the sum of the scores ranges from 0 (the best) to 96 (the worse).
Pain measured with the Numeric Rating Score (NRS) | In rest during intake and in rest and during performance based tests before and after the diagnostic nerve block (if applicable), before the intervention (if applicable), 6 weeks, 3 months, 6 months and 1 year after the intervention
  NRS will be measured in rest and during the performance based tests.
30 seconds chair-stand test | Before and after the diagnostic block, before the intervention (T=0), and at 6 weeks, 3 months, 6 months and 12 months follow up. In the conservative treatment group this will only be done at the applicable follow up dates.
  During this test the total number of complete chair stands (up and down represents one stand) is counted. If at least a full stand is completed at 30 seconds this is counted in the total. If a person cannot stand even once then the score for the test is zero.
40 meters (4x10m) fast-paced walk test | Before and after the diagnostic block, before the intervention (T=0), and at 6 weeks, 3 months, 6 months and 12 months follow up. In the conservative treatment group this will only be done at the applicable follow up dates.
  The total time taken to walk the 4 × 10 m, excluding turns, of one trial is recorded and expressed as speed m/s by dividing distance (40 m) by time (seconds). Timing is paused during turns.
9-steps stair-climb test | Before and after the diagnostic block, before the intervention (T=0), and at 6 weeks, 3 months, 6 months and 12 months follow up. In the conservative treatment group this will only be done at the applicable follow up dates.
  Total time to ascend and descend steps for one trial is recorded in seconds.
Health related quality of life with the EQ-5D-5L | Before the intervention or study start in conservative group (T=0) and during the follow up visits (T=1 at 6weeks, T=2 at 3 months, T=3 at 6 months and T=4 at 12 months after the intervention or study start).
  The EQ-5D descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The respondent is asked to indicate his / her health state by checking the box against the most appropriate statement in each of the five dimensions. EQ-5D comprises a short questionnaire that is cognitively undemanding, taking only a few minutes to complete.
Hospital Anxiety and Depression Scale (HADS) | At T=0 (before intervention) and during T=3 (6 months after intervention)
  The Dutch version of the HADS is a fourteen-item scale with seven items for anxiety (HADS-A) and seven items for depression (HADS-D) (49). Scoring for each item ranges from zero to three. A higher score indicates more anxiety or depression.
Pain Catastrophizing Score (PCS) | At T=0 (before intervention) and during T=3 (6 months after intervention)
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report questionnaire considered to be the most frequent and extensively studied tool to assess pain catastrophizing for chronic pain. Patients are asked to rate the degree to which they have any of the thoughts described in the questionnaire using a 5-point Likert scale ranging from 0 (never) to 4 (always). The total score is the sum of the scores for the individual items, and ranges from 0 to 52. Higher scores indicate a higher level of catastrophizing.
Diagnostic block most appropriate cut-off value | Before and after the diagnostic block and during T=2 (3 months after intervention).
  The continuous results of the diagnostic nerve block in our study (percentage of pain relief) will be used to determine the best cut-off value for the positive outcome of the ablation. The cut-off value will be analysed with a receiver operating curve (ROC) analysis. Results equal or above this cut-off value are considered to predict a positive outcome of the ablation of the nerves, results below the cut-off value are considered to predict a negative outcome of the ablation of the nerve. For this analysis, a positive outcome of the ablation is defined as a MCID in OKS of 4.9 points at 3 months follow up.
Patient satisfaction | During the follow up visits (T=1 at 6weeks, T=2 at 3 months, T=3 at 6 months and T=4 at 12 months after the intervention or study start).
  The patient satisfaction with the result of treatment will be measured with a 5-point Likert scale (1-5). The patients will be asked to grade the statement 'I am satisfied with the result of the treatment' with the following options:
  1. Strongly disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly agree
Patient Global Impression of Change (PGIC) | During the follow up visits (T=1 at 6weeks, T=2 at 3 months, T=3 at 6 months and T=4 at 12 months after the intervention or study start).
  The PGIC in pain and function will be measured with a 5-point Likert scale (1-5) on the applicable follow up visits. The patients will be asked to rate the following statements:
  * Please imagine how you would have described your pain intensity before the procedure. How do you feel today as compared to baseline (Start of the study) as far as your knee pain caused by OA is concerned?
  * Please imagine how you would have described the functionality of your knee before the procedure. How do you feel today as compared to baseline (start of the study) as far as your knee functionality caused by OA is concerned?
  The options on the Likert scale are:
  1. much better
  2. slightly better
  3. no change
  4. slightly worse
  5. much worse
Minimal Clinically Important Difference (MCID) of the OKS | MCIDs will be determined for our population on T=1 (6weeks), T=2 (3 months) and T=3 (6 months) follow up. .
  We will use distribution and anchor based methods to determine the MCID on the patient reported outcomes of the OKS.
Minimal Clinically Important Difference (MCID) of the WOMAC | MCIDs will be determined for our population on T=1 (6weeks), T=2 (3 months) and T=3 (6 months) follow up.
  We will use distribution and anchor based methods to determine the MCID on the patient reported outcomes of the WOMAC.
Minimal Clinically Important Difference (MCID) for the EQ-5D-5L | MCIDs will be determined for our population on T=1 (6weeks), T=2 (3 months) and T=3 (6 months) follow up.
  To determine the MCID on the patient reported outcomes of the EQ-5D-5L we will use an instrument defined method.
Minimal Clinically Important Difference (MCID) of the 30 seconds chair-stand test | MCIDs will be determined for our population on T=1 (6weeks), T=2 (3 months) and T=3 (6 months) follow up.
  We will use distribution and anchor based methods to determine the MCID of the 30 seconds chair-stand test.
Minimal Clinically Important Difference (MCID) of the 40 meters (4x10m) fast-paced walk test | MCIDs will be determined for our population on T=1 (6weeks), T=2 (3 months) and T=3 (6 months) follow up.
  We will use distribution and anchor based methods to determine the MCID of the 40 meters (4x10m) fast-paced walk test.
Minimal Clinically Important Difference (MCID) of the 9-steps stair-climb test. | MCIDs will be determined for our population on T=1 (6weeks), T=2 (3 months) and T=3 (6 months) follow up.
  We will use distribution and anchor based methods to determine the MCID of the 9-steps stair-climb test.
Adverse events | After the diagnostic block, after the intervention (T=0), and at 6 weeks, 3 months, 6 months and 12 months follow up.
  The reported treatment related or probably treatment related adverse events will be listed as numbers with frequencies per treatment.
Medication changes | Before the intervention (T=0), and at 6 weeks, 3 months, 6 months and 12 months follow up.
  The patients will be asked to report changes in the use of NSAIDs and opioids during the follow up visits. The results will be summarised as increased use, no change, decrease in use and use of opioids will be reported as MME.
Number of Total Knee Artroplasty's (TKA's) | At 6 weeks, 3 months, 6 months and 12 months follow up.
  The number of TKAs during the study follow up will be documented including the point in time since the intervention. If applicable, we will use the Kaplan-Meier estimator to estimate the survival function.
Procedure time | During the intervention visit (T=0)
  The total procedure time of chemical ablation and RFA will be measured in minutes. The measurement starts as soon as the treating physician puts on his sterile gloves and will end when the sterile draping is taken off.

CONTACTS AND LOCATIONS:
Overall Officials: Gezina Oei, MD, PhD, Principal Investigator — Academic Medical Centre Amsterdam; Markus Hollmann, Prof, Study Chair — Academic Medical Centre Amsterdam
Locations (2):
- Netherlands (2):
  - Dijklander Ziekenhuis, Hoorn, North Holland
  - Bravis Ziekenhuis, Roosendaal

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and the final data will be published. Conditions for reuse apply: A de-identified dataset will be made available upon request to the corresponding author. The request must include ethics approval and a statistical analysis plan.
  An embargo period applies: The embargo period is at least 1 year after the publication of the original study.
Time Frame: An embargo period applies: The embargo period is at least 1 year after the publication of the original study.
Access Criteria: A de-identified dataset will be made available upon request to the corresponding author. The request must include ethics approval and a statistical analysis plan. Digital data and documentation will be preserved for 15 years.

REFERENCES:
- [Derived] Wit PR, Beek RV, Schokker M, Wensing C, Hollmann MW, Kallewaard JW, Oei G; RADIOPHENOL collaborators; Collaborative group name. Genicular nerve radiofrequency ablation, phenol neurolysis or conservative medical management in patients with knee osteoarthritis: protocol for the RADIOPHENOL randomised controlled multicentre trial with three parallel groups. BMJ Open. 2025 Jul 6;15(7):e094576. doi: 10.1136/bmjopen-2024-094576. PMID 40623740